CLINICAL TRIAL: NCT07067593
Title: Benefits and Risks of Amnioreduction for Management of Pregnant Women With Polyhydramnios
Brief Title: Amnioreduction in Polyhydramnios
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed Gamal M.fekry, Lecturer obstetric and gynecology, Specialist Urogynecology, Assiut University
Other Study IDs: AMN
Record Dates: First submitted 2025-07-06; First posted 2025-07-16 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Polyhydramnios
Keywords: Amnioreduction; Polyhydramnios
MeSH Terms: conditions — Polyhydramnios

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Amnioreduction
- Conservative

SUMMARY:
The aim of this work is to review the indications, procedural complications and outcomes of amnioreduction in pregnancies complicated by polyhydramnios.

DETAILED DESCRIPTION:
Polyhydramnios is the presence of excessive amniotic fluid in the amniotic sac and it's prevalence reaches 2% of all pregnancies . Polyhydramnios is diagnosed based on ultrasound criteria, as an amniotic fluid index (AFI) >25 cm or maximal vertical pocket > 8 cm . There is a recognized association of polyhydramnios and adverse pregnancy outcomes, including perinatal death, fetal abnormality and preterm birth . Management of the pregnancy can be problematic, particularly in severe cases, due to issues surrounding maternal discomfort and the risk of preterm birth. Amnioreduction, widely used in the management of polyhydramnios, is an option available to palliate maternal symptomatology and potentially prolong the pregnancy . Previous publications have shown a reduction in the risk for premature rupture of membranes and preterm labor decrease, placental perfusion improvement, and relief of maternal discomfort following amnioreduction

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women 20- 38 weeks
* Patients with polyhydramnios

Exclusion criteria:

* Lethal fetal anomalies
* Pre labor rupture of membranes
* Placental separation
* Chorioamnionitis

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All pregnant women between 24 to 38 weeks attending Fetal Medicine Unit at Women's health hospital for antenatal care or admitted due to antepartum hemorrhage or for scheduled surgery and meeting the inclusion criteria are counseled to participate in our study after informed consent. sample size will be devided into 2 groups:
  Group 1 : patients with Amnioreduction Group 2 : patients with conservative management (without amnioreduction)
Sampling Method: Non-Probability Sample
Enrollment: 28 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Gestational age at delivery | 4 months
  Determine Gestational age at delivery in polyhydramnios patients . Increased age is good.
Rate of PROM | 4 months
  Number of cases developed PROM

CONTACTS AND LOCATIONS:
Locations (1):
- Women's Health Hospital, Asyut, Egypt